CLINICAL TRIAL: NCT02742701
Title: Comparison of Glycosuria and Capillary Blood Glucose in Hospitalised Diabetic Patients
Brief Title: Diabetes and Palliative Care
Acronym: DIAPAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maison Médicale Jeanne Garnier (Other)
Responsible Party: Sponsor
Other Study IDs: MMJG/2014/SC/001
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: End-of-life; Diabetes; Terminal Cancer
MeSH Terms: conditions — Death; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: diagnosis — Measurement of glycosuria

SUMMARY:
Diabetes prevalence in palliative care is 10-15%. Most hospice patients are treated with insulin. The target glucose level is high in order to decrease the risk of hypoglycemia. Glucose level is usually monitored using capillary blood glucose once to three times daily.

The aim of the research is to simplify this pattern of care in end-of-life patients. It will evaluate whether the non invasive measurement of glucose in urine could replace the measurement of capillary blood glucose. The first objective will be to assess the performance of the measurement of glucosuria using urinary dip stix to predict that the blood glucose level is within the target range.

Due to the high glucose target, hyperglycemia is extremely frequent. However, symptoms of hyperglycemia are unfrequently reported. They may be unspecific and/or masked in end-of-life patients due to terminal disease and medication. The second objective of the study will be to define symptoms of hyperglycemia in these patients.

DETAILED DESCRIPTION:
This is a prospective study involving several palliative care units in France. Glycemia and glycosuria will be measured in the same patients. Symptoms that could be related to hyperglycemia will be assessed in relation with the concomitant blood glucose level.

Main investigations :

Glycosuria and cetonuria will be measured using a dip stix during each nursing care.

Glycemia will be measured before breakfast and before diner. Pain caused by finger pricking for the measurement of glycemia will be evaluated using a verbal scale.

Symptoms will be evaluated at the time of each glucose measurement first with open questions then with a list of potential symptoms of hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients
* hospitalised in a palliative care unit
* terminally ill with cancer
* with blood glucose measurement at least twice daily over 5 days
* agreeing to participate in the study

Exclusion Criteria:

* patient unable to communicate, to understand information about the study or to decline participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in a palliative care unit
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of glycosuria measured on urine collected between 10 am and 16 am on the blood glucose level at 6 pm | over 12 days
  Glycosuria will be assessed using Ketodiabur 5000 urinary dip stix. The results are semi-quantitative with 8 levels of glycosuria ranging from 0% to 2% (weight/volume).
  Capillary blood glucose level will be assessed using a glucose meter based on glucose oxydase.

SECONDARY OUTCOMES:
Relation between glycemia and glycosuria at different time points over 24 hours. | over 12 days
  Glycemia and glycosuria will be assessed as described above.
Intensity of pain caused by finger pricking | 12 days
  Intensity of pain will be assessed using a simple numerical scale.
Type, frequency and intensity of symptoms in relation to the blood glucose level | 12 days
  Intensity of symptoms will be assessed using a simple numerical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Guirimand, MD, Principal Investigator — Pôle Recherche Maison Médicale Jeanne Garnier

IPD SHARING:
Plan to Share IPD: No